CLINICAL TRIAL: NCT04081181
Title: CT_ Guided Percutaneous Microwave Ablation in Treatment of Pulmonary Malignancies
Brief Title: Microwave Ablation in Pulmonary Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Reham M Farghally, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MWAL
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT_ guided percutaneous microwave ablation (Experimental): The procedure will be done under anaesthesia by interventional radiologist
  Interventions: Procedure: Microwave ablation

INTERVENTIONS:
Procedure: Microwave ablation — CT_guided Microwave ablation is a minimally invasive technique that kill the insitu lung cancer cells, produce large volumes of cellular necrosis with reduced procedure time .According to the preoperative CT image of the patient , we will determine the focal position of the lesion ,it's size and it's relationship with adjacent organs to choose the optimal puncture point , puncture path and proper microwave antenna and to set the power and time of ablation.Then under the guidance of CT , the tip of antenna will be sent into the focus by puncture with ablation power of 60_80 W .according to tumor size , the ablation time will be determined.Needle track coagulation will be done to prevent seeding of malignant cells. After ablation a CT scan will be done immediately to observe the size ,shape and relation to nearby organ of the lesion and to determine if there is pneumothorax

SUMMARY:
Lung cancer remains to be an important global issue as it is the leading cause of cancer_ related mortality for both men and women worldwide .Since more than two thirds of cases are diagnosed at an advanced stage,the survival rate of lung cancer is one of the lowest among all cancers.

DETAILED DESCRIPTION:
Currently , Surgery is one of the curative treatment option for primary lung cancer but most patients are either diagnosed at an advanced stage or are unfit for surgery due to medical co_morbidities or poor underlying lung reserve , less than a third of all lung cancer patients can undergo surgical resection .

Lung metastasectomy is considered a therapeutic option increasing the survival rate for patients of pulmonary metastases but only 25%_30% of patients benefits from lung metastasectomy due to multiplicity of pulmonary nodules or medical co_ morbidities .

In spite of a significant improvement of lung cancer chemotherapy and radiotherapy in recent years , the overall clinical outcome is less than satisfactory compared with that brought by surgical resection .Thus , it is urgent to provide a method which is more effective than chemotherapy and radiotherapy and nearly effective as the surgical treatment for the patients who are not eligible for surgery.

Local thermal ablation therapy of the tumor is the focus of recent research in the past decades .This method is to deliver specific energy into the tumor tissue under the guidance of image technology , which make the local tissue quickly reach 60°C where an irreversible coagulative necrosis happens leading to necrosis of tumor cells .

CT_guided Microwave ablation is a minimally invasive technique that may be an alternative treatment option for management of lung cancer in patients who are not candidate for surgery .This method not only kill the insitu lung cancer cells , but also protect lung cancer tissue .It can produce large volumes of cellular necrosis with reduced procedure time , can use multiple antennae and can be used in lesions with cystic component and/or in proximity to vascular structures.

Thus, CT guided microwave ablation is a promising new technique that is convenient ,easy ,causing less trauma ,associated with no need for general anaesthesia , fast recovery and less complications.

ELIGIBILITY:
Inclusion Criteria:

* patient has good compliance and sign the informed consent.

  * patient with lung cancer who lost the opportunity of surgical resection.
  * patient has one or more metastatic lung nodules (not more than 5)

Exclusion Criteria:

* patient is pregnant or breast feeding .

  * patient with uncorrectable coagulopathy.
  * There are large blood vessels or important structures adjacent to lung lesion.
  * patient with more than five nodules

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2020-07-15 (Estimated); Primary Completion 2022-05-13 (Estimated); Study Completion 2022-08-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients achieving adequacy of ablation | 24 hours post ablation
  Defined as perilesional circumferential solid area of ground glass opacification of >4mm
Percentage of patients achieving technical efficacy | 1 month after ablation
  Defined as lack of enhancement within the ablated zone
Local progression free survival | From the date of ablation up to six months
  The interval between microwave ablation and evidence of local recurrence. Local recurrence defined as enlargement of the zone , the development of contrast enhancement in the part of the zone or change in the size of the ablated zone as a result if enlargement of one area.

SECONDARY OUTCOMES:
Adverse events | From the date of ablation up to six months follow up
  Defined as incidence of intra , peri and post procedural complications

REFERENCES:
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Jahangeer S, Forde P, Soden D, Hinchion J. Review of current thermal ablation treatment for lung cancer and the potential of electrochemotherapy as a means for treatment of lung tumours. Cancer Treat Rev. 2013 Dec;39(8):862-71. doi: 10.1016/j.ctrv.2013.03.007. Epub 2013 Apr 17. PMID 23601905
- [Background] Weiser MR, Downey RJ, Leung DH, Brennan MF. Repeat resection of pulmonary metastases in patients with soft-tissue sarcoma. J Am Coll Surg. 2000 Aug;191(2):184-90; discussion 190-1. doi: 10.1016/s1072-7515(00)00306-9. PMID 10945362
- [Background] Smith R, Pak Y, Kraybill W, Kane JM 3rd. Factors associated with actual long-term survival following soft tissue sarcoma pulmonary metastasectomy. Eur J Surg Oncol. 2009 Apr;35(4):356-61. doi: 10.1016/j.ejso.2008.01.004. Epub 2008 Feb 21. PMID 18294807
- [Background] Zhong L, Sun S, Shi J, Cao F, Han X, Bao X, You Q. Clinical analysis on 113 patients with lung cancer treated by percutaneous CT-guided microwave ablation. J Thorac Dis. 2017 Mar;9(3):590-597. doi: 10.21037/jtd.2017.03.14. PMID 28449467
- [Background] Bonichon F, Godbert Y, Gangi A, Buy X, Palussiere J. PET/Computed Tomography and Thermoablation (Radiofrequency, Microwave, Cryotherapy, Laser Interstitial Thermal Therapy). PET Clin. 2015 Oct;10(4):519-40. doi: 10.1016/j.cpet.2015.05.008. Epub 2015 Aug 1. PMID 26384598
- [Background] Shahzad Y, Louw R, Gerber M, du Plessis J. Breaching the skin barrier through temperature modulations. J Control Release. 2015 Mar 28;202:1-13. doi: 10.1016/j.jconrel.2015.01.019. Epub 2015 Jan 20. PMID 25616160
- [Background] Simon CJ, Dupuy DE, Mayo-Smith WW. Microwave ablation: principles and applications. Radiographics. 2005 Oct;25 Suppl 1:S69-83. doi: 10.1148/rg.25si055501. PMID 16227498
- [Background] Carrafiello G, Lagana D, Mangini M, Fontana F, Dionigi G, Boni L, Rovera F, Cuffari S, Fugazzola C. Microwave tumors ablation: principles, clinical applications and review of preliminary experiences. Int J Surg. 2008;6 Suppl 1:S65-9. doi: 10.1016/j.ijsu.2008.12.028. Epub 2008 Dec 14. PMID 19186116
- [Background] Cheng M, Fay M, Steinke K. Percutaneous CT-guided thermal ablation as salvage therapy for recurrent non-small cell lung cancer after external beam radiotherapy: A retrospective study. Int J Hyperthermia. 2016 May;32(3):316-23. doi: 10.3109/02656736.2015.1137640. Epub 2016 Feb 19. PMID 26892261
- [Background] Pacella CM, Papini E. Image-guided percutaneous ablation therapies for local recurrences of thyroid tumors. J Endocrinol Invest. 2013 Jan;36(1):61-70. doi: 10.1007/BF03346744. PMID 23391859
- [Background] Anderson EM, Lees WR, Gillams AR. Early indicators of treatment success after percutaneous radiofrequency of pulmonary tumors. Cardiovasc Intervent Radiol. 2009 May;32(3):478-83. doi: 10.1007/s00270-008-9482-6. Epub 2009 Jan 6. PMID 19127381
- [Background] Chheang S, Abtin F, Guteirrez A, Genshaft S, Suh R. Imaging Features following Thermal Ablation of Lung Malignancies. Semin Intervent Radiol. 2013 Jun;30(2):157-68. doi: 10.1055/s-0033-1342957. PMID 24436532